CLINICAL TRIAL: NCT06714071
Title: Relation of C-reactive Protein/ Albumin Ratio and Coagulation Profile in Acute Myeloid Leukemia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, shrouk mosallam ahmed khalaf, doctor, Assiut University
Other Study IDs: aml and crp/albumin ratio
Record Dates: First submitted 2024-11-08; First posted 2024-12-03 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: AML
MeSH Terms: interventions — Bleeding Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CRP and Albumin and coagulation profile — CRP and Albumin and coagulation profile

SUMMARY:
The investigators will investigate the relation between CAR and coagulation profile in newly diagnosed AMl patients

DETAILED DESCRIPTION:
Acute myeloid leukaemia (AML) is an aggressive haematological malignancy with a high degree of heterogeneity. It has long been recognized that systemic inflammation is associated with tumorigenesis it revealed that elevated C-reactive protein levels were associated with worse survival outcomes in patients with various types of cancer, including hematologic malignancies. Serum albumin is a measure of an individual's nutritional status. Systemic inflammation can reduce serum albumin concentrations by increasing capillary permeability . The ratio of CRP to albumin (CAR) is a useful score based on inflammation and nutrition, reflecting not only systemic inflammation status but also nutritional status. The Glasgow prognostic score (GPS) and modified GPS (mGPS), determined by the serum CRP and albumin levels, have been proposed as prognostic indicators for AML patients. However, the clinical correlations of CAR and its prognostic value in AML patients have not yet been clarified. Abnormalities of hemostasis can occur in leukemia in the form of disseminated intravascular coagulation(DIC), coagulation protein defect and primary fibrinolysis . Clinically, Types of acute myeloid leukemia like acute promyelocyticleukemia has a high frequency of haemorrhage due to disseminated intravascular coagulation (DIC), which contributes to the high mortality rate of this disease . Therefore, the investigators will investigate CAR its relation with inflammatory response and coagulation profile levels in newly diagnosed acute myeloid leukemia and after 3 month follow up to compare their level and the relation between .

ELIGIBILITY:
Inclusion Criteria:

- all cases newly diagnosed with acute myeloid leukemiain assuit university hospital

Exclusion Criteria:

1. cases with chronic myeloid leukemia
2. cases with acute lymphoblasticleukemia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all cases newly diagnosed with acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between C- reactive protein and coagulation profile in AML patients | Study complete an average 2 years
  the investigators will investigate the correlation between CAR and coagulation profile in newly diagnosed AMl patients by measure crp and coagulation profile in newly diagnosed patient and up to 3 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: sohir kamel, prof, Study Director — Director
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided